CLINICAL TRIAL: NCT00044681
Title: A Study to Evaluate the Efficacy, Safety and Maintenance Effect of Risperidone Augmentation of SSRI Monotherapy in Young and Older Adult Patients With Unipolar Treatment-Resistant Depression
Brief Title: A Study of the Effectiveness and Safety of Risperidone to Augment SSRI Therapy in Patients With Treatment-resistant Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002143
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-11

CONDITIONS: Depressive Disorder; Depressive Disorder, Major; Depression
Keywords: Risperidone; depression; melancholia; depressive disorder; antipsychotic agents
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of risperidone to augment SSRI therapy in patients with treatment-resistant depression and to demonstrate the long-term maintenance effect of risperidone as augmentation therapy compared with placebo augmentation in these patients.

DETAILED DESCRIPTION:
Treatment strategies for treatment-resistant depression (TRD) involve either switching to another antidepressant, augmenting the first-line treatment with various pharmacologic agents, or switching to a different medication in combination with another agent. This study includes 2 phases: an open-label treatment phase and a double-blind maintenance phase, during which neither the patient nor the physician knows whether risperidone or placebo is administered. The open-label phase has an initial period of 6 weeks during which patients with TRD receive only citalopram, a selective serotonin reuptake inhibitor (SSRI). Risperidone is then added to the treatment regimen for 4 weeks to evaluate its short-term effect in augmenting the therapy. The double-blind phase last for 6 months and evaluates the relapse prevention of continued risperidone augmentation therapy compared with placebo augmentation of the SSRI. Targeted daily doses of citalopram and risperidone are adjusted for younger adults (18 to 54 years of age) and older adults (55 to 85 years of age). Assessments of effectiveness include the Montgomery-Asberg Depression Rating Scale (MADRS); Hamilton Rating Scale of Depression (HAM-D); Clinical Global Impression of Severity (CGI-S); response rate, determined by the proportion of patients showing >=50% improvement on MADRS total score; and relapse, evaluated by changes in CGI or HAM-D scores. Safety evaluations include the incidence of adverse events throughout the study, vital signs (pulse and blood pressure) and weight, and clinical laboratory tests (hematology, biochemistry, urinalysis) at specified intervals. The study hypothesis is that risperidone augmentation of SSRI therapy will show significant improvement in symptoms of depression compared with SSRI monotherapy and that risperidone augmentation will show better time-to-relapse than placebo augmentation in patients with TRD. Once daily, oral tablets of risperidone (0.25 milligram[mg], 0.5mg, 1.0mg, and 2.0mg), citalopram (20mg and 40mg) or placebo. Risperidone for 30 weeks; 0.25-2.0mg for younger adults, 0.25-1.0mg for older adults. Citalopram for 36 weeks; 20-60 mg for younger adults; 20-40 mg for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria of Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV), for Major Depressive Disorder
* history of resistance to therapy with antidepressant medication
* score on the Hamilton Rating Scale of Depression (HAM-D) of >=20 at start of study.

Exclusion Criteria:

* Meet DSM-IV criteria for Axis I disorder (except anxiety disorders) or borderline personality disorder
* substance dependence, including drugs of abuse and alcohol
* history of schizophrenia, bipolar disorder, or manic episode
* meet DSM-IV criteria for delirium, dementia, amnesic or other cognitive disorder supported by Mini Mental Status Examination (MMSE)
* pregnant or nursing females, or those lacking adequate contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2002-10; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score at end of treatment; time to relapse

SECONDARY OUTCOMES:
Response rate, determined from >=50% improvement from baseline at MADRS total score; change from baseline in Hamilton Rating Scale of Depression (HAM-D) and Clinical Global Impression (CGI) scale; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study to Evaluate the Efficacy, Safety and Maintenance Effect of Risperidone Augmentation of SSRI Monotherapy in Young and Older Adult Patients with Unipolar Treatment-Resistant Depression — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=451&filename=CR002143_CSR.pdf